CLINICAL TRIAL: NCT02888574
Title: Evaluating the Efficacy of Intranasal Oxytocin Among Individuals With Persistent Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Tavis S. Campbell, Professor, University of Calgary
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CHREB16-0334
Record Dates: First submitted 2016-08-30; First posted 2016-09-05 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Chronic Pain; Pelvic Pain
MeSH Terms: conditions — Chronic Pain; Pelvic Pain | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intranasal Oxytocin (Experimental): Oxytocin nasal spray delivered bi-daily over a 14-day period at 24-IU per dose
  Interventions: Drug: Intranasal Oxytocin
- Placebo (Placebo Comparator): Placebo nasal spray containing the same ingredients as the active nasal spray minus the oxytocin and packaged in an identical bottle. To be delivered bi-daily over a 14-day period at 24-IU per dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intranasal Oxytocin — Intranasal oxytocin (Syntocinon; Novartis, Switzerland)
  Other Names: Syntocinon
  Arms: Intranasal Oxytocin
Drug: Placebo — Placebo nasal spray
  Arms: Placebo

SUMMARY:
This study is a placebo-controlled, double-blind, within-participants crossover investigation of the effect of intranasal oxytocin on pain and function among women with chronic pelvic pain.

DETAILED DESCRIPTION:
1. Rationale: Oxytocin (OT) is a neuropeptide produced in the supraoptic and paraventricular nuclei of the hypothalamus. There exists at least three plausible mechanisms through which OT may decrease pain sensitivity. In brief, the first mechanism involves spinal signaling. A direct hypothalamo-spinal projection originating from the paraventricular nucleus transports OT, to the dorsal horn (Lamina-I, II, and IV), an area containing OT receptors that influence glutamate and GABA cellular signaling. The second mechanism involves an indirect pathway via the endogenous opioids. Evidence suggests that OT binds to opioid receptors and may also stimulate endogenous opioid release in the brain. Finally, OT may decrease pain by improving mood, decreasing anxiety, and mitigating the stress response.

   Thirty-three animal investigations have assessed OT-pain relationships with 29 reporting that exogenous administration and higher endogenous levels decreased pain. There is a lack of clarity of an OT-pain association in the human literature due to a paucity of methodologically rigorous trials. Thus far, OT administration has been reported to lower pain sensitivity among patients experiencing chronic back pain, headache, constipation, and colon pain. To date, no research has evaluated the association between intranasal OT and chronic pelvic pain. The association between OT and pain may be different in women with pelvic pain relative to other chronic pain conditions because of a potential peripheral OT-pain pathway. There is an abundance of OT receptors in the uterus, and OT is a potent uterogenic agent that is clinically used in large doses to stimulate uterine contractions and induce labor. While OT does not cross the blood-brain-barrier, the central administration of intranasal OT increases central and blood-plasma OT concentrations. Thus, intranasal OT administration may be associated with pain through central and peripheral pathways; however uterine contractions with 24IU doses of intranasal OT occur in only 1 in every 100-1000 people.
2. Research questions and objectives: This research is a pilot study of the efficacy of intranasal OT at improving pain and function among women with chronic pelvic pain of primarily musculoskeletal origin.
3. Design: This study will utilize a double-blind, placebo-controlled, within-subjects crossover design. Participants will complete 6-weeks of testing consisting of two 2-week intranasal administrations separated by a 2-week washout period

ELIGIBILITY:
Inclusion Criteria:

* Non-menopausal women with chronic pelvic musculoskeletal pain (i.e., pain exceeding 6-months in duration that is located primarily in the pelvic region and reproducible on palpation to the muscles spanning the pelvic floor) will be eligible to participate if they: 1) have regular menstrual periods (monthly within a 21-35 day range); 2) using a permanent or barrier form of contraception; 3) can commit not to change their medication during the 6-weeks of this study; and 4) have a moderate amount of pain at baseline (i.e., a pain score of 4-7 out of 10 on a numeric rating scale). A baseline pain score of 4-7 out of 10 was selected to prevent floor and ceiling effects and ensure that participants have room to change throughout the course of the study.

Exclusion Criteria:

* Muscle pain as a result of systemic disease, scoring positive on a urine pregnancy test, concurrent use of another nasal spray, nasal pathology (e.g., ears, nose, and throat diagnosis), diabetes insipidus, previous or concurrent use of narcotics delivered intranasally (e.g., cocaine), are contemplating pregnancy, or who have sacroiliac instability as defined by the European Guidelines. Women will also be excluded with they have a primary diagnosis of endometriosis, dysmenorrhea, interstitial cystitis, functional bowel disorder, fibromyalgia or neuropathic pain.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Self-reported pain | 14-days
  The Brief Pain Inventory - Short Form

SECONDARY OUTCOMES:
Self-report positive and negative affect | 14-days
  Positive and Negative Affect Scale
Self-report depressed mood, anxious mood, and stress | 14-day
  Depression Anxiety Stress Scale
Self-report sleep | 14-day
  Medical Outcomes Study Sleep Scale

CONTACTS AND LOCATIONS:
Overall Officials: Tavis S Campbell, PhD, Principal Investigator — University of Calgary
Locations (1):
- Behavioural Medicine Laboratory, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Flynn MJ, Campbell TS, Robert M, Nasr-Esfahani M, Rash JA. Intranasal oxytocin as a treatment for chronic pelvic pain: A randomized controlled feasibility study. Int J Gynaecol Obstet. 2021 Mar;152(3):425-432. doi: 10.1002/ijgo.13441. Epub 2020 Dec 8. PMID 33112417
- [Derived] Rash JA, Toivonen K, Robert M, Nasr-Esfahani M, Jarrell JF, Campbell TS. Protocol for a placebo-controlled, within-participants crossover trial evaluating the efficacy of intranasal oxytocin to improve pain and function among women with chronic pelvic musculoskeletal pain. BMJ Open. 2017 Apr 16;7(4):e014909. doi: 10.1136/bmjopen-2016-014909. PMID 28416501